CLINICAL TRIAL: NCT01914016
Title: Functional Electrical Stimulation for People With Multiple Sclerosis Who Experience Foot Drop:Feasibility of Instrumented Gait Analysis in Clinical Practice.
Brief Title: Functional Electrical Stimulation for People With Multiple Sclerosis Who Experience Foot Drop
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Margaret University (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Principal Investigator, Marietta van der Linden, Senior Research Fellow, Queen Margaret University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: QMU ELHF109-121
Record Dates: First submitted 2013-06-25; First posted 2013-08-01 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- prolonged walk (Other)
  Interventions: Other: prolonged walk

INTERVENTIONS:
Other: prolonged walk — Participants will be asked to walk for a duration of between 2 -6 minutes until they rate their perceived exertion as 'Hard' (RPE 16 on Borg Scale)

SUMMARY:
People with Multiple Sclerosis (pwMS) often experience 'foot-drop' which means that the foot is not adequately lifted during the so-called swing phase (foot is off the ground) during walking which can lead to trips and falls. Functional Electrical Stimulation (FES) to the shin muscles will aid lifting of the foot and therefore reduces the risk of trips and falls. There have been several studies showing the benefits of FES to the walking of pwMS. The proposed study aims to optimise the FES prescription and fitting care pathway for pwMS in Edinburgh and the Lothians This will be achieved firstly through a survey to all clients with MS in the last 5 years who have been regarded as suitable for FES. Secondly, a pilot study will assess the suitability of the use of simple clinical measurement (electrogoniometry) which will allow the measurement of the degree of foot-drop. The degree is foot drop is usually assessed by the physiotherapist using visual observation. Using a small device which can be quickly fitted to the patient's lower and foot for the duration of a 2-6 minute walk, the physiotherapist will be able to quantify the degree of foot drop over time. Such a measurement is especially important for people with MS who are often affected by increased mental and physical fatigue.

Our first hypothesis is that the degree of foot-drop at the end of the walk is increased compared to the start of the walk. Secondly, we hypothesise that the degree of foot drop is less when the participant walks with the assistance of Functional Electrical Stimulation at their next clinical appointment.

DETAILED DESCRIPTION:
Participants People with MS (aged 18 or over) who are assessed for their suitability for FES to treat foot-drop at Slateford Medical Centre are eligible for participation in this study.

For this feasibility study we aim to recruit at least 10 participants.

Recruitment Eligible patients will be given an information sheet by their physiotherapist who will introduce the study at their initial appointment. A second appointment is made to fit the FES unit and if the patient is willing to consider taking part in the study, informed consent is taken.

Data collection To record the degree of foot-drop, one arm of the electrogoniometer will be attached to the side of the participant's lower leg and the other arm to the shoe using skin-friendly double sided adhesive tape.

The participant will then be asked to walk in their normal walking speed around the corridors of the clinic for six minutes or shorter if the participant is not able to walk for this duration. A data logger carried on the belt on the participant's waist will continuously record the ankle angle data at 50Hz. Walking speed will be derived by measuring the distance walked in the time recorded. Rate of perceived exertion on the Borg Scale will be recorded every minute and immediately after the walk. Participants will also be asked to fill in a questionnaire on their perceived walking performance (Multiple Sclerosis Walking Scale 12).

At a follow-up appointment (1-2 weeks later) this data collection will be repeated with the participant using the FES unit.

Data analysis. To assess the impact of fatigue on the ankle angle during prolonged walking, ankle angle data in the first and last 60 seconds of the walk will be recorded. Two way ANOVA will be employed to analyse both the effects of time (within session) and that of FES use ('Off' and 'On', between sessions) on the degree of foot-drop if data are normally distributed. Equivalent non-parametric statistics will be used for non normally distributed data. Statistical significance will be accepted at p<0.05.

Inclusion criteria People with MS (aged 18-80) who are assessed for their suitability for FES to treat foot-drop between September 2013 and March 2014 at Slateford Medical Centre are eligible for participation in this study.

Exclusion criteria Patients with fixed ankle deformities, who are allergic to tape and who are unable to walk for at least for two minutes (with or without walking aids) will be excluded. Patients who experienced a relapse or any trauma affecting their walking between the first fitting appointment and the follow-up appointment will also be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* People with MS (aged 18-80) who are assessed for their suitability for FES to treat foot-drop between September 2013 and March 2014 at Slateford Medical Centre are eligible for participation in this study

Exclusion Criteria:

* Patients with fixed ankle deformities, who are allergic to tape and who are unable to walk for at least for two minutes (with or without walking aids) will be excluded.
* Patients who experienced a relapse or any trauma affecting their walking between the first fitting appointment and the follow-up appointment will also be excluded from the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-09; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Peak dorsiflexion angle during the swing phase without FES | Baseline
  The electrogoniometer record the (sagittal) ankle angle during the 2-6 minute walk around the physiotherapy department. In the data processing stage, the peak dorsiflexion angle during the swing phase will be determined for each gait cycle over a period of 20 seconds at the start and at the end of the walk.

SECONDARY OUTCOMES:
Rate of perceived exertion (RPE) | Baseline
  The participant will be asked to rate his/her perceived exertion on the Borg Scale (6-20) at minute intervals during the walk.
Peak dorsiflexion angle during swing phase (with FES) | two weeks from baseline
  The electrogoniometer record the (sagittal) ankle angle during the 2-6 minute walk around the physiotherapy department. In the data processing stage, the peak dorsiflexion angle during the swing phase will be determined for each gait cycle over a period of 20 seconds at the start and at the end of the walk.
Rates of perceived Exertion (RPE) with FES | 2 weeks from baseline
  The participant will be asked to rate his/her perceived exertion on the Borg Scale (6-20) at minute intervals during the walk

OTHER OUTCOMES:
MS walking scale | baseline and 2 weeks from baseline
  The participant will be asked to fill in the MS walking scale, for both without (first visit) and with walking with the assistance of FES (second visit) in mind.

CONTACTS AND LOCATIONS:
Overall Officials: Marietta L van der Linden, PhD, Principal Investigator — Queen Margaret University
Locations (1):
- Slateford medical centre, Edinburgh, United Kingdom